CLINICAL TRIAL: NCT04247438
Title: Polysaccharide-based, Artificial Biofilm Substitute - Clinical Pilot Study for Validation Process
Brief Title: Dentures Biofilm and Artificial Biofilm Substitute
Acronym: KÜBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TUDKW20200115; 427547277 (Other Grant/Funding Number: German Research Foundation (DFG))
Record Dates: First submitted 2020-01-13; First posted 2020-01-30 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Biofilm
Keywords: dental biofilm; dental plaque; polysaccharides; chitosan; methylcellulose; denture biofilm; denture plaque; biofilm model
MeSH Terms: conditions — Dental Plaque | interventions — Dentures

STUDY DESIGN:
Intervention Model Description: Single group, prospective, longitudinal, interventional pilot study to test the feasibility of study design, protocol, and methods for evaluating the artificial dentures biofilm equivalent. This pilot study is intended to provide initial data and insights into the development and establishment of an artificial dentures biofilm equivalent. According to the current state of research, no data, therefore, are available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biofilm formation (Other): Biofilm formation after 12 and 36 h on PMMA (polymethyl methacrylate) dentures and the number of brushing cycles needed to remove it.
  Interventions: Other: 12h and 36h Biofilm formation on PMMA (Palapress®) dentures and samples worn by participants and brushing cycles needed to remove it.

INTERVENTIONS:
Other: 12h and 36h Biofilm formation on PMMA (Palapress®) dentures and samples worn by participants and brushing cycles needed to remove it. — Capturing the clinical data for biofilm formation on PMMA dentures and samples worn by participants and the number of brushing cycles required to remove this biofilm.
  Development of artificial denture biofilm substitute with similar mechanical properties to real denture biofilm.

SUMMARY:
The biofilm on oral surfaces can lead to oral diseases. The correlation between oral biofilm and diseases and general health is well known. Therefore, cleaning of teeth or dentures from biofilm is essential for the maintenance of oral and general health. Currently, the society is ageing, the number of elderly as well as home and institutionalized care patients is increasing. In particular, these suffer from higher tooth loss, wear removable dentures and have problems with independent oral and denture hygiene. Therefore, support from well-trained nursing staff or family members is important. The use of suitable artificial biofilm substitutes may be helpful, in order to efficiently and easily perform oral and denture hygiene education, as well as to carry out laboratory tests of oral and denture hygiene products. The absence of such appropriate substitutes for denture biofilm requires innovations in this field. The aim of this pilot study is to verify the feasibility of the study protocol, design and methods. Additionally, an innovative artificial biofilm substitute based on polysaccharides will be further developed. This pilot study includes five study parts. Two in vivo examinations and three in vitro tests. This pilot study creates the basis for further main studies and implements the development of validated artificial biofilm substitutes.

DETAILED DESCRIPTION:
The bacterial biofilm on the intraoral surfaces is a three-dimensionally structured, firmly adhering layer of microorganisms surrounded by a matrix of extracellular polymeric substances (EPS). This matrix can take up to 90% of the biofilm mass. Biofilm on oral surfaces can lead to diseases such as caries, periodontitis or denture stomatitis. Furthermore, an association between denture biofilm, which serves as a reservoir for various bacteria, and general diseases is described. Adequate denture hygiene is therefore essential for maintaining the health of denture wearers. Nevertheless, adequate oral and denture hygiene is not sufficiently available for many, especially institutionalized elderly. The reasons are mostly insufficient preventive measures to train denture wearers, nursing staff and family members, as well as a lack of training materials such as dentures with artificial biofilm equivalents, which have the same cleaning properties as real dentures biofilm.

The absence of such appropriate substitutes for denture biofilm requires innovations in this field. Further, clinical data for validation of innovative artificial biofilm substitutes are missing.

The aim of this pilot study is to carry out preliminary tests for the development of a polysaccharide-based artificial biofilm substitute to simulate the real denture biofilm and to verify the feasibility of the study protocol, design and methods i.e. recording the obligatory manual and mechanical brushing cycles or for adapting the mechanical properties and adhesive strength to the clinically recorded data.

This pilot study includes 2 in vivo and 3 in vitro parts. The in vivo examinations contain 8 visits for participants. For biofilm formation participants omit cleaning dentures for 12 and 36 hours. Biofilm formation occurs between the visits and removal within the visits. Digital planimetry will be performed to measure the biofilm formation and removal. Within 3 in vitro tests, the mechanical properties of the artificial biofilm substitutes will be adjusted and the reliability tested. The artificial biofilm contains chitosan and methylcellulose. The mechanical brushing cycles needed to remove artificial biofilm substitutes, will be measured by a tooth-brushing simulator under standardized conditions. Digital planimetry of artificial biofilm after brushing will be performed.

The collected data will be used for further conceptualization of the main study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older
* Individuals wearing sufficient acrylic resin (PMMA) complete upper or complete upper and lower denture
* healthy oral mucosa
* written informed consent

Exclusion Criteria:

* Individuals who have severe systemic and/or infectious diseases
* Female individuals who are pregnant or breastfeeding
* allergies or hypersensitivity to the used products and/or materials
* smokers
* Individuals with a history of chronic drug abuse or another illness which does not allow the participant to assess the nature and/or possible consequences of the study
* inability to comply with study protocol requirements
* Individuals who have participated in another clinical study less than 4 weeks prior to the baseline examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
dentures brushing cycles 12 h in vivo | 2 days
  Capturing the data for the number of brushing cycles needed to remove artificial biofilm from dentures worn by participants for 12h.
brushing cycles in vitro | 4 months
  Capturing the data for the number of brushing cycles needed to remove artificial biofilm from dentures or samples.

SECONDARY OUTCOMES:
percentage of plaque (POP) | 3 - 12 weeks
  Measuring of denture area covered with biofilm by digital planimetry.
dentures brushing cycles 36 h in vivo | 4 days
  Capturing the data for the number of brushing cycles needed to remove artificial biofilm from dentures worn by participants for 36 h.
samples brushing cycles 12 h in vivo | 2 days
  Capturing the data for the number of brushing cycles needed to remove artificial biofilm from samples worn by participants for 12h.
samples brushing cycles 36 h in vivo | 4 days
  Capturing the data for the number of brushing cycles needed to remove artificial biofilm from samples worn by participants for 36 h.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Walczak, Dr.med.dent., Study Chair — Department of Prosthetik Dentistry, Faculty of Medicine, TU Dresden
Locations (1):
- Department of Prosthetic Dentistry, Carl Gustav Carus Faculty of Medicine, TU Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen WH, Burne RA, Wu H, Koo H. Oral Biofilms: Pathogens, Matrix, and Polymicrobial Interactions in Microenvironments. Trends Microbiol. 2018 Mar;26(3):229-242. doi: 10.1016/j.tim.2017.09.008. Epub 2017 Oct 30. PMID 29097091
- [Background] Flemming HC, Wingender J. The biofilm matrix. Nat Rev Microbiol. 2010 Sep;8(9):623-33. doi: 10.1038/nrmicro2415. Epub 2010 Aug 2. PMID 20676145
- [Background] Nikawa H, Hamada T, Yamamoto T. Denture plaque--past and recent concerns. J Dent. 1998 May;26(4):299-304. doi: 10.1016/s0300-5712(97)00026-2. PMID 9611934
- [Background] Coulthwaite L, Verran J. Potential pathogenic aspects of denture plaque. Br J Biomed Sci. 2007;64(4):180-9. doi: 10.1080/09674845.2007.11732784. PMID 18236742
- [Background] Russell SL, Boylan RJ, Kaslick RS, Scannapieco FA, Katz RV. Respiratory pathogen colonization of the dental plaque of institutionalized elders. Spec Care Dentist. 1999 May-Jun;19(3):128-34. doi: 10.1111/j.1754-4505.1999.tb01413.x. PMID 10860077
- [Background] El-Solh AA, Pietrantoni C, Bhat A, Okada M, Zambon J, Aquilina A, Berbary E. Colonization of dental plaques: a reservoir of respiratory pathogens for hospital-acquired pneumonia in institutionalized elders. Chest. 2004 Nov;126(5):1575-82. doi: 10.1378/chest.126.5.1575. PMID 15539730
- [Background] Hoad-Reddick G, Grant AA, Griffiths CS. Investigation into the cleanliness of dentures in an elderly population. J Prosthet Dent. 1990 Jul;64(1):48-52. doi: 10.1016/0022-3913(90)90152-3. PMID 2384898